CLINICAL TRIAL: NCT04120675
Title: The Effects of Early Harvest Extra Virgin Olive Oil on Cognition and Mental Health of Primary (PPMS) or Secondary (SPMS) Progressive Multiple Sclerosis Patients
Brief Title: Efficacy of Early Harvest Olive Oil in Cognition of Primary (PPMS) or Secondary (SPMS) Progressive Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Greek Alzheimer's Association and Related Disorders (Other); Ellis-Farm, Eliama Daily Value Gold (ellis-farm.com) (Unknown)
Responsible Party: Principal Investigator, Magda Tsolaki, MD, PhD, Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43-Α/24-10-2018
Record Dates: First submitted 2019-09-24; First posted 2019-10-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Progressive Multiple Sclerosis
Keywords: extra virgin olive oil; cognition; mental health; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Psychological Well-Being; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental Group 20 patients on Early Harvest Extra Virgin Olive Oil Aluminum bottle with 500 ml of early harvest extra virgin olive oil (3 tablespoons per day).
  Dietary Supplement: Early Harvest Extra Virgin Olive Oil dietary intake of the content of 50 mL (3 tablespoons from the bottle containing the product)
  Interventions: Dietary Supplement: Early Harvest Extra Virgin Olive Oil
- Control group (Active Comparator): 10 patients will not receive treatment with Extra Virgin Olive Oil
  Interventions: Dietary Supplement: Early Harvest Extra Virgin Olive Oil

INTERVENTIONS:
Dietary Supplement: Early Harvest Extra Virgin Olive Oil — Participants will take 3 tablespoons on a daily basis

SUMMARY:
To date, no drug therapy has been approved for primary (PPMS) & secondary (SPMS) progressive multiple sclerosis. The urgent need to find new therapies - if possible with minimal side effects - led us to the search for the potential therapeutic effects of early harvest olive oil. The positive effect of phenol-rich, flavonoid and lignin-based olive oil on the modification of intestinal microbe populations and their by-products of metabolism is well known, such as the extent of gut-associated lymphoid tissue immune-stimulation due to antioxidants, anti-inflammatory and immunoregulatory properties. The aim of this Greek, Randomized Clinical Trial, is to evaluate the effect of Early Harvest Extra Virgin Olive Oil on cognition and mental health of patients diagnosed with PPMS or SPMS. The patients will be evaluated once at the beginning of treatment, after 6 months of treatment and after twelve months of treatment, in order to specify the eficacy of extra virgin olive oil in holistic treatments for SPMS and PPMS

DETAILED DESCRIPTION:
Study Type: Randomized Clinical Trial. Primary Purpose: Prevention OBJECTIVES OF THE TRIAL The objectives of this study are:To investigate the efficacy of Early Harvest EVOO as a disease course modifying treatment for primary (PPMS) or secondary (SPMS) progressive multiple sclerosis in a phase III randomized controlled clinical trial study in objective measurements in patients with primary (PPMS) or secondary (SPMS) progressive multiple sclerosis.

STUDY DESIGN This is a Greek, randomized controlled study group of Early Harvest EVOO to a control group, in which the patients will receive only their symptomatic medication. Qualifying patients will be randomly assigned to receive 50mL of Early Harvest EVOO or not on a daily basis for 24 months. Patients undergo assessments at baseline, 6 and 12 months +/- 7 days after beginning treatment.

Duration: The total study duration will be 12 months. Patients will receive study interventions for 12 months.

Number of Subjects 30 subjects total will be enrolled; 20 in the experimental group (Early Harvest EVOO); 10 in the Control group

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary (PPMS) or secondary (SPMS) progressive multiple sclerosis
* EDSS≥ 5
* No response to any given treatment for MS or interruption due to side effects
* Progressive aggravation in the disease's progression estimated by: deterioration in EDSS-plus disability scale, Timed 25-Foot Walk or 9-hole peg test.
* Progressive aggravation in the disease's progression estimated by: new lesions in MRI scan and neuropsychological tests
* Progressive aggravation in patient's neuropsychological status
* Progressive aggravation in patient's Quality of life, estimated with MuSIQol - Greek 3.01 MS and SF-36
* Years of education: >= 5
* Proficient language fluency
* Have a study partner with 10+ hr/wk contact (can be in person and telephone), accompanies to visits
* Compliance

Exclusion Criteria:

* Enrollment in other trials or studies not compatible with MSOIL
* Visual and auditory acuity inadequate for neuropsychological testing
* History of significant other neurological or psychiatric illnesses or presence of other diseases precluding enrollment.
* Use of forbidden medications (listed below)
* Ferromagnetic implants and devices (including implants or devices held in place by sutures, granulation or ingrowth of tissue, fixation devices, or by other means) not eligible for MRI scanning. Brain malformation or other conditions that may complicate lumbar puncture
* Any significant or uncontrolled medical condition or treatment-emergent
* Clinically significant laboratory abnormality

Medications across the study

Excluded Medication:

* Immunosuppressant or immunomodulating agents, corticosteroids, or investigational drugs within 3 months of study initiation
* Antibiotics in general, at least one month prior assessment of specific inflammatory markers (faecal levels of calprotectin, metabolomic profile, gut microbiota)
* Use of neuroleptics or within 4 weeks of screening
* Participation in any other investigational drug study within 4 weeks of screening (individuals may not participate in any drug study while participating in this protocol).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
Greek Verbal Learning Test (GVLT)- Assessment of auditory and verbal memory | baseline, 6 and 12 months
  Changes in Greek Verbal Learning Test (GVLT) score. Score range:0-80. Higher score indicates better outcome
Brief Visuospatial Memory Test (BVMT)- Assessment of visual and spatial memory | baseline, 6 and 12 months
  Changes in Brief Visuospatial Memory Test (BVMT) score. Score range:0-36. Higher score indicates better outcome
Symbol Digit Modalities Test (SDMT)- Assessment of processing speed and working memory | baseline, 6 and 12 months
  Changes in Symbol Digit Modalities Test (SDMT) score. Score range:1-110. Higher score indicates better outcome
Perceived Deficits Questionnaire (PDQ)- Measurement of subjective cognitive deficits | baseline, 12 and 24 months
  Changes in Perceived Deficits Questionnaire (PDQ) score. Score range:0-80. Lower score indicates better outcome
Frontal Assessment Battery (FAB)- Assessment of frontal deficits | baseline, 6 and 12 months
  Changes in Frontal Assessment Battery (FAB) score. Score Range:0-18. Higher score indictaes better outcome
Beck Depression Scale (BDI)- Measurement of depressive symptoms | baseline, 6 and 12 months
  Changes in Beck Depression Scale (BDI) score. Score range:0-63. Lower scores indicate better outcomes.
Mental Health Inventory (MHI)- Measurement of emotional condition and mental health problems | baseline, 6 and 12 months
  Changes in Mental Health Inventory (MHI) score. Score range:0-100. Higher score indicates better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- A' Department of Neurology,Aristotle University of Thessaloniki (AUTH), Thessaloniki, Macedonia, Greece

IPD SHARING:
Plan to Share IPD: Undecided